CLINICAL TRIAL: NCT06389929
Title: Do the Health Education Materials Developed in the Gynecology and Diseases Nursing Course Affect Students' Teaching Material Motivation and Material Design Self-Efficacy Beliefs?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Simge Ozturk, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IU-HB-RK-02
Record Dates: First submitted 2024-01-28; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Nursing Caries
Keywords: nursing; Gynecological health and disease nursing; Health education material,; Teaching material motivation; Material design self-efficacy belief
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled n = 86 (43 = control, 43 = intervention) students who took the Women's Health and Diseases Nursing course at Bartın University, Faculty of Health Sciences, Department of Nursing and volunteered to participate in the study were randomly assigned to two groups: intervention and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skill Group (Experimental): Students in the skill group will take one of the applications in the Skill Checklists (Breastfeeding Education Skill Check Form, Breast Care and Caregiving to Mothers with Breast Engorgement Skill Check Form, Breast Self-Examination (KKMM) Training Skill Check Form) within the scope of the "Women's Health and Diseases Nursing Course". Health education material was prepared in line with the skills they determined. The duration of training material preparation is determined as 1 week for each student. The health education material developed was prepared and presented by evaluating the reason, importance, awareness aspect and innovative perspective of the determined skill.
  Interventions: Behavioral: Education
- Control Group (No Intervention): The post-test will be applied to the control group 1 day after the pre-test, and the questionnaires and scales applied in the pre-test to the skill group were re-evaluated after the presentation of the health education material.

INTERVENTIONS:
Behavioral: Education — In line with the skill they will determine for one of the applications in the Skill Checklists (Breastfeeding Education Skill Control Form, Breast Care and Giving Care to Mothers with Breast Engorgement Skill Control Form, Breast Self-Examination (KKMM) Training Skill Control Form) apply.
  Arms: Skill Group

SUMMARY:
Purpose: This study aimed to examine the effect of health education material developed by nursing students in gynecological health and disease nursing on students' teaching material motivation and material design self-efficacy belief.

Method: The study was conducted as a prospective randomized controlled study. n=86 (43=control, 43=intervention) students who took the Women's Health and Diseases Nursing course at Bartın University Faculty of Health Sciences Nursing Department between 30.10.2023-20.01.2024 and volunteered to participate in the study were randomized. It was conducted in two groups: intervention and control.In the research, data will be collected with the Data Collection Form prepared by reviewing the literature, Instructional Material Motivation Scale and Material Design Self-Efficacy Belief Scale. Descriptive statistics, Student t-test, Mann-Whitney U Test, Wilcoxon Signed Rank Test and Pearson correlation tests will be used to evaluate the data.

DETAILED DESCRIPTION:
Aim: This study aimed to examine the effect of health education material developed by nursing students in women's health and disease nursing on students' teaching material motivation and material design self-efficacy beliefs.

Method: The study was conducted as a prospective randomized controlled study. n=86 (43=control, 43=intervention) students who took the Women's Health and Diseases Nursing course at Bartın University Faculty of Health Sciences Nursing Department between 30.10.2023-20.01.2024 and volunteered to participate in the study were randomized. It was conducted in two groups: intervention and control. In the research, data will be collected with the Data Collection Form prepared by reviewing the literature, Instructional Material Motivation Scale and Material Design Self-Efficacy Belief Scale. Descriptive statistics, Student t-test, Mann-Whitney U Test, Wilcoxon Signed Rank Test and Pearson correlation tests will be used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Students who were over 18 years old,
* Students who spoke Turkish,
* Students who were not diagnosed with hearing impairment,
* Students who took the Gynecology and Diseases Nursing course,
* Students who had written consent
* Students who volunteered to participate

Exclusion Criteria:

* Not studying at Bartın University,
* students who did not take the Gynecology and Diseases Nursing course

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Instructional Material Motivation Scale | two weeks
  The original version of the scale was published by Keller (2010). PMSQ, a 36-item measurement tool consisting of five-point Likert type options (not true, somewhat true, true, moderately true, very true), was developed by taking the ARCS Model as a criterion. The measurement tool consists of four sub-dimensions with the same name as the compliance, trust, satisfaction and attention components of the ARCS Model. The 3rd, 7th, 12th, 15th, 19th, 22nd, 29th, 31st and 34th items of the measurement tool have negative expressions and require reverse scoring. The lowest score that can be obtained from the measurement tool, whose midpoint is 108.00, is 36.00, while the highest score is 180.00 (Keller, 2010).
  Increasing scores from the scale indicate an increase in motivation. The original version of the scale was applied to university students by Keller (2006), and as a result of the analyzes made for the sub-dimensions of the measurement tool.

SECONDARY OUTCOMES:
Material Design Self-Efficacy Belief Scale | two weeks
  In order to determine material design self-efficacy beliefs, the Material Design Self-Efficacy Belief Scale developed by Bakaç and Özen (2015) was used. The validity and reliability study of the scale was conducted on 300 teacher candidates who studied at Abant İzzet Baysal University in the 2013-2014 academic year and had previously taken the ÖTMT course. The construct validity of the scale was tested by exploratory and confirmatory factor analysis, and a scale with three dimensions (Material Preparation on Computer, Three-Dimensional Material Design and Two-Dimensional Material Design) and 25 items was created, explaining 48% of the total variance. The scale items are 5-point Likert type and are as follows: "Strongly Disagree", "Disagree", Undecided", Agree" and "Strongly Agree".
  Increasing scores from the scale indicate an increase in motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Simge OZTURK, Bartın, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No